CLINICAL TRIAL: NCT00895141
Title: Changes in LDL and HDL With Increased Intake of Saturated Fat From Dairy Foods in Individuals With Atherogenic Dyslipidemia and LDL Subclass Pattern B
Brief Title: Effect of Saturated Fat on Large Low-density Lipoprotein (LDL) and High-density Lipoprotein (HDL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: Dairy Management Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MM3355
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Dyslipidemia
Keywords: Saturated fat; LDL size; Large LDL; Large HDL
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low saturated fat diet (Experimental): Moderate carbohydrate (35%E), moderate protein (25%E), high fat (40%E) diet with 8%E saturated fat
  Interventions: Dietary Supplement: Saturated Fat Diet
- High saturated fat diet (Experimental): Moderate carbohydrate (35%E), moderate protein (25%E), high fat (40%E) diet with 20%E saturated fat
  Interventions: Dietary Supplement: Saturated Fat Diet

INTERVENTIONS:
Dietary Supplement: Saturated Fat Diet — Moderate carbohydrate (35%E), moderate protein (25%E), high fat diet (40%E) with 8%E saturated fat
  Arms: Low saturated fat diet
Dietary Supplement: Saturated Fat Diet — Moderate carbohydrate (35%E), moderate protein (25%E), high fat (40%E) diet with 20%E saturated fat
  Arms: High saturated fat diet

SUMMARY:
The purpose of the study is to test whether increased saturated fat intake results in increased levels of larger LDL and HDL particles in individuals with LDL Pattern B.

DETAILED DESCRIPTION:
Increased saturated fat intake is known to elevate plasma levels of both low-density lipoprotein cholesterol (LDL-C) and high-density lipoprotein cholesterol (HDL-C), however, less is know regarding the effect of saturated fat on lipoprotein subclasses. We previously showed that, in the context of a reduced carbohydrate diet, saturated fat induced increases in LDL cholesterol were apparently due to increases in large, more buoyant LDL without increases in small, dense LDL. This finding was supported by a previous dietary intervention study showing a correlation between saturated fat intake and large LDL. In both cases, this increase in large LDL was correlated with an increase in large HDL. In this study, we will test the following specific hypotheses regarding changes in plasma lipoproteins induced by a diet high in myristic acid and other saturated fats derived primarily from dairy sources in individuals with LDL subclass pattern B: 1) there will be a coordinate increase in levels of large HDL particles that are considered anti-atherogenic and large LDL particles that are less strongly associated with increased CVD risk than smaller LDL; 2) this change in lipoprotein profile will result in a higher proportion of pattern B individuals converting to LDL subclass pattern A (predominance of larger LDL); and 3) the coordinate increase in large HDL and LDL is due to a common underlying pathway. The latter hypothesis will be addressed by assaying cholesterol ester transfer protein (CETP), hepatic lipase (HL), and lipoprotein lipase (LPL).

ELIGIBILITY:
Inclusion Criteria:

* Men or postmenopausal woman between 18-70 yrs
* Body Mass Index between 25-35
* Blood pressure <150/90
* Non smoking
* Agrees to consume no alcohol or dietary supplements during the study
* LDL Subclass Pattern B
* Total cholesterol and LDLC ≤95th percentile for sex and age
* Fasting triglycerides ≤ 500mg/dl
* Fasting blood sugar < 126 mg/dl
* At least 3 months weight stable

Exclusion Criteria:

* History of coronary heart disease, cerebrovascular disease, peripheral vascular disease, bleeding disorder, liver or renal disease, diabetes, lung disease, HIV, or cancer (other than skin) in the last 5 years
* Taking drugs known to affect lipid metabolism or hormones
* Abnormal thyroid stimulating hormone (TSH)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-04; Primary Completion 2010-09 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Large LDL (LDL I + 2a) (mg/dl) | 3 wk, 6 wk
Large HDL (HDL2b) (mg/dl) | 3 wk, 6 wk
LDL peak particle size | 3 wk, 6 wk

SECONDARY OUTCOMES:
Triglycerides (mg/dl) | 3 wk, 6 wk
Total Cholesterol (mg/dl) | 3 wk, 6 wk
LDL cholesterol (mg/dl) | 3 wk, 6 wk
HDL cholesterol (mg/dl) | 3 wk, 6 wk
Apolipoprotein AI (mg/dl) | 3 wk, 6 wk
Apolipoprotein B (mg/dl) | 3 wk, 6 wk
Medium LDL (LDL2b) (mg/dl) | 3 wk, 6 wk
Small LDL (LDL3a) (mg/dl) | 3 wk, 6 wk
Hepatic Lipase Activity | 3 wk, 6 wk
Lipoprotein Lipase Activity | 3 wk, 6 wk
Cholesteryl Ester Transfer Protein Activity | 3 wk, 6 wk
Very Small LDL (LDL3b, 4a, 4b) (mg/dl) | 3 wk, 6 wk

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Krauss, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- Cholesterol Research Center, Berkeley, California, United States

REFERENCES:
- [Derived] Chiu S, Williams PT, Krauss RM. Effects of a very high saturated fat diet on LDL particles in adults with atherogenic dyslipidemia: A randomized controlled trial. PLoS One. 2017 Feb 6;12(2):e0170664. doi: 10.1371/journal.pone.0170664. eCollection 2017. PMID 28166253